CLINICAL TRIAL: NCT03358745
Title: Impact of Meal Order on Postprandial Cardiometabolic Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Vinnova (Other Government); Anti-Diabetic Food Centre (Other)
Responsible Party: Principal Investigator, Juscelino Tovar, Project Leader, Lund University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AFC2016-17.JT
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Metabolic Syndrome X; Insulin Resistance; Hyperinsulinism; Glucose Metabolism Disorders; Metabolic Diseases
Keywords: Type 2 diabetes risk; Cardiovascular disease risk
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Hyperinsulinism; Glucose Metabolism Disorders; Metabolic Diseases | interventions — Bread; Butter; Cheese; Salads

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard meal, bread/butter as starter (Experimental): Subjects eat a reference lunch (reference lunch) at 11:30 am, 4 h after a defined light breakfast. The meal contains 38 g fat and 885 kcal and consists of bread and butter, soup, salad and cheese. The participants eat the bread and butter portion within 15 min and the remaining components of the meal are consumed within the following 15 min (total eating time=30 min).
  Blood samples are taken before the lunch and every 30 min postprandial for 4 h.
  Interventions: Other: Standard meal, bread/butter as starter
- Standard meal with soup as starter (Experimental): Subjects eat a reference lunch (reference lunch) at 11:30 am, 4 h after a defined light breakfast. The meal contains 38 g fat and 885 kcal. The participants eat the soup portion within 15 min and the remaining components of the meal are consumed within the following 15 min (total eating time=30 min).
  Interventions: Other: Standard meal with soup as starter
- Standard meal with cheese as starter (Experimental): Subjects eat a reference lunch (reference lunch) at 11:30 am, 4 h after a defined light breakfast. The meal contains 38 g fat and 885 kcal. The participants eat the cheese portion within 15 min and the remaining components of the meal are consumed within the following 15 min (total eating time=30 min).
  Interventions: Other: Standard meal with cheese as starter
- Standard meal with salad as starter (Experimental): Subjects eat a reference lunch (reference lunch) at 11:30 am, 4 h after a defined light breakfast. The meal contains 38 g fat and 885 kcal. The participants eat the salad portion within 15 min and the remaining components of the meal are consumed within the following 15 min (total eating time=30 min).
  Interventions: Other: Standard meal with salad as starter

INTERVENTIONS:
Other: Standard meal, bread/butter as starter — Reference lunch. Bread and butter are eaten during the first 15 min. Soup, cheese and salad are eaten within the following 15 min.
  Arms: Standard meal, bread/butter as starter
Other: Standard meal with soup as starter — Lunch meal in which soup is eaten during the first 15 min. Bread, butter, cheese and salad are eaten within the following 15 min.
  Arms: Standard meal with soup as starter
Other: Standard meal with cheese as starter — Lunch meal in which cheese is eaten during the first 15 min. Bread, butter, soup and salad are eaten within the following 15 min.
  Arms: Standard meal with cheese as starter
Other: Standard meal with salad as starter — Lunch meal in which salad is eaten during the first 15 min. Bread, butter, soup and cheese are eaten within the following 15 min.
  Arms: Standard meal with salad as starter

SUMMARY:
The order in which the different components of a meal are eaten may have impact on the postprandial metabolic responses to carbohydrates, fat and proteins. This study will compare blood lipids and glycemia regulation following lunches of identical composition but varying the order of intake of the different meal components.

DETAILED DESCRIPTION:
The order in which the different components of a meal are eaten may have impact on the postprandial metabolic responses to carbohydrates, fat and proteins. Some of these responses are associated with the risk for developing cardiometabolic complications.

The study will be carried out in a cohort of healthy subjects with a wide BMI range and normal fasting glycemia. Postprandial metabolic responses to a reference meal starting with bread and butter (BB) will be compared with those registered after 3 other meals of identical composition, in which the starter will be permutated. Each meal is tested on an independent experimental session, with a 1 week washout interval.

The intervention will be carried out at the Food for Health Science Centre - Lund University. Additionally, the plan contemplates an initial information visit including screening of fasting blood glucose. In total, each volunteer completing the study will pay five visits to the clinical unit.

Based on the results from the above-described phase, a second step of the study will compare various quality attributes of the most effective starter on the impact on cardiometabolic risk markers, as a way to optimize putative protective actions and to gain further mechanistic insight.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 30 kg/m2
* Fasting blood glucose ≤ 6.1 mmol/L
* No known medical condition

Exclusion Criteria:

* Smoking habits
* Treatment for high blood pressure
* Treatment for hypercholesterolemia

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve of postprandial glycemia | 4 hours postprandial
  Area under the curve of postprandial glycemia (0-4h) after each intervention, compared to the reference meal.
  Plasma glucose is measured pre-meal and and at various post-meal intervals for up to for 4 hours. AUC is calculated and compared to AUC recorded after the reference meal.

SECONDARY OUTCOMES:
Area under the curve (AUC) of postprandial triglyceridemia | 4 hours postprandial
  Area under the curve (AUC) of postprandial triglyceridemia (0-4h) after each intervention, compared to the reference meal
Area under the curve (AUC) of postprandial insulinemia | 4 hours postprandial
  Area under the curve (AUC) of postprandial insulinemia (0-4h) after each intervention, compared to the reference meal
Area under the curve (AUC) of postprandial Glucagon-like peptide (GLP-1), Peptide YY (PYY) and glucose-dependent insulinotropic polypeptide (GIP) | 4 hours
  Area under the curve (AUC) of postprandial GLP-1, GIP and PYY (0-4h) after each intervention, compared to the reference meal

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Antidiabetic Food Centre, Chemical Centre. Lund University, Lund, Skåne County
  - Food for Health Science Centre. Lund University Medicon Village, Lund

REFERENCES:
- [Background] Jakubowicz D, Wainstein J, Ahren B, Bar-Dayan Y, Landau Z, Rabinovitz HR, Froy O. High-energy breakfast with low-energy dinner decreases overall daily hyperglycaemia in type 2 diabetic patients: a randomised clinical trial. Diabetologia. 2015 May;58(5):912-9. doi: 10.1007/s00125-015-3524-9. Epub 2015 Mar 1. PMID 25724569
- [Background] Esquirol Y, Bongard V, Mabile L, Jonnier B, Soulat JM, Perret B. Shift work and metabolic syndrome: respective impacts of job strain, physical activity, and dietary rhythms. Chronobiol Int. 2009 Apr;26(3):544-59. doi: 10.1080/07420520902821176. PMID 19360495
- [Background] Lee SH, Tura A, Mari A, Ko SH, Kwon HS, Song KH, Yoon KH, Lee KW, Ahn YB. Potentiation of the early-phase insulin response by a prior meal contributes to the second-meal phenomenon in type 2 diabetes. Am J Physiol Endocrinol Metab. 2011 Nov;301(5):E984-90. doi: 10.1152/ajpendo.00244.2011. Epub 2011 Aug 9. PMID 21828339
- [Background] Dejeans N, Herosimczyk A, Sayd T, Chambon C, Martin JF, Maier JA, Tauveron I, Mazur A. Effect of a high-fat challenge on the proteome of human postprandial plasma. Clin Nutr. 2013 Jun;32(3):468-71. doi: 10.1016/j.clnu.2012.05.017. Epub 2012 Jun 19. PMID 22721722